CLINICAL TRIAL: NCT03966209
Title: Evaluation of PD-1 Inhibition in Patients With Recurrent Hepatocellular Carcinoma After Liver Transplantations
Brief Title: Safety and Efficacy of PD-1 Inhibitors in Patients With Liver Transplant
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Principal Investigator, Jian Zhou, Professor, Shanghai Zhongshan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JS001LT
Record Dates: First submitted 2019-05-27; First posted 2019-05-29 (Actual); Last update posted 2019-05-31 (Actual); Status verified 2019-05

CONDITIONS: Hepatocellular Carcinoma; Liver Transplantation
Keywords: Checkpoint Inhibitor; Immunotherapy
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment (Experimental): JS001（PD-1 inhibitor）, 240mg I.V. Q3W,
  Interventions: Drug: JS001(PD-1 inhibitor)

INTERVENTIONS:
Drug: JS001(PD-1 inhibitor) — 240mg I.V. Q3W

SUMMARY:
This is a perspective clinical study to assess the safety and efficacy of PD-1 inhibitors in patients with LT. Eligible patients have recurrent or metastatic cancer after LT, are not amenable to, or refractory after, locoregional therapy or to a curative treatment approach (eg, surgery, or ablation) and have previously been treated with sorafenib or other targeted therapy, either intolerant to this treatment or show radiographic progression after treatment.

Biopsy is needed to exclude patients with positive allograft PD-L1 expression.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with recurrence or metastases Hepatocellular carcinoma after liver transplantation that not suitable for surgical resection and Local treatments such as radiofrequency ablation, transcatheter arterial embolization and radiotherapy, been treated with sorafenib or other targeted therapy and are either intolerant to this treatment or show radiographic progression after treatment.
2. Age 18-70 years old, male or female
3. Biopsy shows negative allograft PD-L1 expression
4. Child-Pugh score ≤ 6 points (Child-Pugh A)
5. Estimated postoperative survival time ≥ 12 weeks
6. ECOG score 0-1 points
7. Laboratory test indicators: white blood cells ≥ 3.0 × 109 / L, platelets ≥ 80 × 109 / L, hemoglobin ≥ 100g / L; total bilirubin ≤ 2.5 times the upper limit of normal, transaminase (AST, ALT) ≤ 2.5 times Upper limit of normal value, serum creatinine ≤ 1.5 times normal upper limit
8. Have sufficient understanding and voluntarily sign informed consent to participate in clinical research

Exclusion Criteria:

1. Biopsy shows positive allograft PD-L1 expression
2. Severe allergic reactions to other monoclonal antibodies
3. Have any history of active autoimmune diseases or autoimmune diseases
4. The presence of active infection with Hepatitis B or Hepatitis C Virus
5. Severe cardiopulmonary dysfunction patients, have high blood pressure and blood pressure can not be controlled with drugs, unstable coronary artery disease (uncontrollable arrhythmia, unstable angina), non-compensatory congestive heart failure, within 6 months Myocardial infarction

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2021-04-30 (Estimated); Study Completion 2022-10-31 (Estimated)

PRIMARY OUTCOMES:
Serious Adverse Event Rate | 1.5 years
  the occurrence rate of serious adverse event after PD-1 inhibitor treatment
Acute Graft Rejection Rate | 1.5 years
  the occurrence rate of acute graft rejection after PD-1 inhibitor treatment

SECONDARY OUTCOMES:
Objective Response Rate | 3 years
  Objective Response Rate after PD-1 inhibitor treatment
Progression Free Survival Rate | 3 years
  survival time after PD-1 inhibitor treatment till tumor progression
Over all survival Rate | 3 years
  survival time after PD-1 inhibitor treatment till patient death

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Zhongshan Hospital, Shanghai, Shanghai Municipality, China